CLINICAL TRIAL: NCT02890017
Title: Medico-economical Evaluation of Patient-hotel in Urology
Acronym: HOTELAMBU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCl15_ 0513
Record Dates: First submitted 2016-08-24; First posted 2016-09-07 (Estimated); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Surgery for Sacral Nerve Neurostimulation; Surgery for Urinary Artificial Sphincter; Surgery for Prosthetic Penile Implant
Keywords: outpatient surgery; urology medico-economic; hotel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hotel-Ambu (Experimental): Outpatient surgery with a patient-hotel night
  Interventions: Other: postoperative hotel
- conventional hospitalization (Other): conventional hospitalization
  Interventions: Other: conventional hospitalization

INTERVENTIONS:
Other: postoperative hotel — Outpatient surgery First night stay in a defined patient-hotel Patient come for consultation the next morning of surgery to remove the catheter and/or the compressive bandage. The absence of adverse events is checked, the discharge is confirmed and the evaluation questionnaire is given to the patient.
  Postoperative consultation at 1 and 3 months.
  Arms: Hotel-Ambu
Other: conventional hospitalization — Hospitalization for surgery and first postoperative night stay. Postoperative consultation at 1 and 3 months
  Arms: conventional hospitalization

SUMMARY:
This is a medico-economic study of outpatient surgery paired with a night stay in a patient-hotel, compared with a conventional hospitalization for three types of urological surgeries.

The aim is to show that those two strategies are not different in term of adverse effects or rehospitalization, and that the patient-hotel provide a better quality of life at a reduced cost, in order to generate savings for the paying agent: the Healthcare insurance.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Healthcare insurance affiliation
* Surgeries : sacral nerve neurostimulation, urinary artificial sphincter, or prosthetic penile implant
* ASA (American Society of Anesthesiology) score between I and III
* Patients that can be accompanied by a person with a car
* Prior Informed Consent procedure form signed
* Hospitalisation in Lyon Sud Hospital

Exclusion Criteria:

* Refusal of participation or signing the consent form, guardianship or curatorship patients
* Inability to understand the procedure
* History of cognitive or psychiatric disorders
* Non eligibility to out patient
* Pregnant or breastfeeding patients
* No affiliation to Healthcare insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
ICER = Incremental Cost-Effectiveness Ratio of Costs and QALY(quality-adjusted life year) (unit of measure = cost(€)/QALY) | at 3 months
  Efficacity (QALY) is a composite measure of quality of life and adverse events occurence:
  * Quality of life is a composite score of : EQS5D questionnaire converted in utility, Other questionnaires : SF-12 ; International Continence Society short form, Post-Operative Patient, Global Impression of Improvement (PGI-I), l'Incontinence Impact Questionnaire-Short Form (IIQ-SF) et l'Urogenital Distress Index (UDI-SF).
  * Adverse events occurrence : urinary retention, postoperative infection, rehospitalization
  Costs :
  according to " micro-costing " method. Rehospitalizations will be priced from ENC rate.

SECONDARY OUTCOMES:
postoperative complications | at 3 months
  All postoperative complications that occur within 3 months
Change in general quality of life postoperatively measured by EQ5D questionnaire | at Baseline and after surgery at day one
Change in general quality of life postoperatively measured by SF12 questionnaire | at Baseline and after surgery at day one
Change in general quality of life at 3 months after surgery measured by EQ5D questionnaire | at Baseline and at 3 moths
Change in general quality of life at 3 months after surgery measured by SF12 questionnaire | at Baseline and at 3 moths
Change in specific quality of life measured by questionnaires International Continence Society short form | at Baseline and after surgery at day one
Change in specific quality of life measured by Post-Operative Patient questionnaire | at Baseline and after surgery at day one
Change in specific quality of life measured by Global Impression of Improvement (PGI-I) questionnaire | at Baseline and after surgery at day one
Change in specific quality of life measured by Incontinence Impact Questionnaire-Short Form (IIQ-SF) | at Baseline and after surgery at day one
Change in specific quality of life measured by Urogenital Distress Index (UDI-SF) questionnaire | at Baseline and after surgery at day one
Change in specific quality of life measured by International Continence Society short form | at Baseline and at 3 months
Change in specific quality of life measured by Post-Operative Patient questionnaire | at Baseline and at 3 months
Change in specific quality of life measured by Global Impression of Improvement (PGI-I) questionnaire | at Baseline and at 3 months
Change in specific quality of life measured by Incontinence Impact Questionnaire-Short Form (IIQ-SF) | at Baseline and at 3 months
Change in specific quality of life measured by Urogenital Distress Index (UDI-SF) questionnaire | at Baseline and at 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Urologie du Centre Hospitalier Lyon Sud, Hospices Civils de Lyon, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No